

Title: A Phase 1/2, Randomized, Observer-Blind, Placebo-Controlled Trial to Evaluate the Safety and Immunogenicity of TAK-919 by Intramuscular Injection in Healthy Japanese Male and Female Adults Aged 20 Years and Older

NCT Number: NCT04677660

Statistical analysis plan Approve Date: 19-Mar-2021

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black bar) to protect either personally identifiable information or company confidential information.



### STATISTICAL ANALYSIS PLAN

Study Number: TAK-919-1501

licable Terms of Use Study Title: A Phase 1/2, Randomized, Observer-Blind, Placebo-Controlled Trial to Evaluate the Safety and Immunogenicity of TAK-919 by Intramuscular Injection in Healthy Japanese Male and Female Adults Aged 20 Years and Older Version: 1. 0
Date: 19-Mar-2021

Prepared by:

Based on:

Protocol Version: Original Protocol Date: 18Nov2020

### CONFIDENTIAL PROPERTY OF TAKEDA

This document is a confidential communication of Takeda. Acceptance of this document constitutes the agreement by the recipient that no information contained herein will be published or disclosed without written authorization from Takeda.

## **REVISION HISTORY**

| Version | Approval Date | Primary Rationale for Revision | - (5 |
|---------|---------------|--------------------------------|------|
| 1.0 | | [Not Applicable] | Λω. |

Property of Takeda. For noncommercial use only and subject to the applicable

# TABLE OF CONTENTS

| 1 0 | | ODIE | | | | _ |
|---|---|---|---|---|---|---|
| 1.0 | | | | ES, ENDPOINTS AND ESTIMANDS | | |
| | 1.1 | | | es | | |
| | | 1.1.1 | Prıı | mary Objective | | 1 |
| | | 1.1.2 | Sec | ondary Objective(s) | | 7 |
| | | 1.1.3 | Exp | bloratory Objectives | | 7 |
| | 1.2 | Er | ndpoin | ts | | 8 |
| | | 1.2.1 | Pri | nary Endpoint(s) | | 8 |
| | | 1.2.2 | Sec | ondary Objective(s) | | 8 |
| | | 1.2.3 | Exp | ploratory Endpoint(s) | <b>,</b> | 8 |
| 2.0 | | STUD | Y DE | SIGN | | 9 |
| 3.0 | | STAT | ISTIC | AL HYPOTHESES AND DECISION RULES | 1 | ( |
| | 3.1 | St | atistica | ıl Hypotheses | 1 | ( |
| | 3.2 | St | atistica | al Decision Rules | 1 | ( |
| | 3.3 | M | ultiplic | city Adjustment | 1 | ( |
| 4.0 | | SAMI | PLE-S | ZE DETERMINATION | 1 | ( |
| 5.0 | | ANAI | LYSIS | ALTITOTHESES AND DECISION ROEDS | 1 | 1 |
| | 5.1 | <b>A</b> 1 | 1 Scree | ened Subjects Analysis Set | 1 | 1 |
| | 5.2 | Sa | fety A | nalysis Setlysis Set | 1 | 1 |
| | 5.3 | Fu | ıll Ana | lysis Set | 1 | 1 |
| | 5.4 | Pe | r-Prote | ocol Analysis Set | 1 | 1 |
| 6.0 | | | | AL ANALYSIS | | |
| | 6.1 | G | eneral | Considerations | 1 | 2 |
| | | 6.1.1 | | ndling of Treatment Misallocations | | |
| | 6.2 | Di | | on of Subjects | | |
| | 6.3 | | - | aphic and Other Baseline Characteristics | | |
| | | | | nographics | | |
| | | | | dical History and Concurrent Medical Conditions | | |
| | 6.4 | | | on History and Concomitant Medications | | |
| K | 6.5 | | | Analysis (Immunogenicity Analysis) | | |
| 0, | , | 6.5.1 | - | nary Endpoint(s) Analysis | | |
| ) | | | 5.1.1 | Derivation of Endpoint(s) | | |
| | | | 5.1.2 | Main Analytical Approach | | |
| | | 6.5.2 | | ondary Endpoint(s) Analysis | | |
| | | | 5.2.1 | Derivation of Endpoint(s) | | |
| | | · · · | 1 | ~ | | • |

| | 6.5.2 | 2.2 | Main Analytical Approach | 16 |
|---|---|---|---|---|
| | 6.5.3 | Expl | loratory Endpoints Analysis | 17 |
| | 6.5.3 | 3.1 | Derivation of Endpoint(s) | 17 |
| | 6.5.3 | 3.2 | Main Analytical Approach | 218 |
| | 6.5.3 | 3.3 | Assessment of the potential relationship between serum bAb antibody | |
| | | | against SARS-CoV-2 and serum nAb antibody against SARS-CoV-2 | 18 |
| | 6.5.4 | Subg | group Analyses | 18 |
| 6.6 | Safe | ty An | nalysis | 18 |
| | 6.6.1 | Adv | erse Events | 19 |
| | 6.6. | 1.1 | All Adverse Events | 19 |
| | 6.6.2 | Prim | nary Safety Endpoints | 19 |
| | 6.6.2 | | Occurrence of Solicited AEs for 7 Days Following Each Vaccination | |
| | 6.6.2 | | Occurrence of Unsolicited AEs for 28 Days After Each Vaccination | |
| | 6.6.2 | _ | Occurrence of Serious AEs Until Day 57 | |
| | 6.6.2 | | Occurrence of Medically-Attended Adverse Events Until Day 57 | |
| | 6.6.2 | - | AEs Leading to Discontinuation of Vaccination | |
| | 6.6.2 | - | AEs Leading to Subject's Withdrawal From the Trial Until Day 57 | |
| | 6.6.2 | | SARS-CoV-2 Infection Until Day 57. | |
| | 6.6.3 | | ondary safety endpoints | |
| | 6.6.3 | | Occurrence of Serious AEs Throughout the Trial | |
| | 6.6.3 | | Occurrence of MAAEs Throughout the Trial | 23 |
| | 6.6.3 | 3.3 | AEs Leading to Subject's Withdrawal From the Trial From the Day of Vaccination Throughout the Trial | 23 |
| | 6.6.3 | 3.4 | This analysis will be conducted only at the Final analysis. SARS-CoV- | |
| | | < | 2 Infection Throughout the Trial | |
| | 6.6.4 | . ( ) , | r Adverse Event Safety Endpoint | |
| | 6.6.4 | | Adverse Events with an Outcome of Death throughout the trial | |
| | 6.6.4 | | Unsolicited Adverse Events of Hypersensitivity | |
| | 6.6.4 | | Related Unsolicited Adverse Events of Hypersensitivity | |
| く、 | 6.6.5 | | er Safety Analysis | |
| | 6.6.5 | | Laboratory Evaluations | |
| | 6.6.5 | | Vital Sign Measurements | |
| | 6.6.6 | Exte | ent of Exposure and Compliance | |
| | 6.6.6 | 5.1 | Exposure to Study Intervention | |
| | 6.6.6 | | Compliance with Study Intervention | |
| | 6.6.7 | Subg | group Analyses | 26 |

| TAK-919-1501<br>Statistical Analys | sis Plan 1.0 | <br>19-Mar-2021 |
|---|---|---|
| 6.7 Inte | rim Analyses | 26 |
| 70 REFER | FNCFS | 27 |
| 8.0 CHANG | GES TO PROTOCOL PLANNED ANALYSES | 27 |
| 9.0 APPEN | IDIX | 28 |
| | inges From the Previous Version of the SAP | |
| 9.2.1 | a Handling ConventionsGeneral Data Reporting Conventions | 28 |
| 9.2. | | 28 |
| 9.2.2 | Definition of Baseline | 30 |
| 9.2.3 | Definition of Baseline | 30 |
| 9.2.4 | Definition of Visit Windows | 30 |
| 9.2.5 | Tables for Laboratory and Vital Sign Abnormalities | 31 |
| 9.2.6 | Tables for Unsolicited Adverse Events of Hypersensitivity | 34 |
| 9.3 Pro | gramming Conventions for Output | 44 |
| 9.4 Ana | ılysis Software | 46 |
| Table 6.a Solic | TEXT TABLES ited Local (Injection Site) Reactions and Systemic AEss the Clinical Safety Laboratory Tests | 20 |
| Table 9.a Anal | ysis Windows for Immunogenicity by Visit | |
| LIST OF IN-T | TEXT FIGURES | |
| Figure 2.a Scho | ematic of Trial Design | 10 |
| Figure 2.a School | | |

### **ABBREVIATIONS**

AE adverse event

ATC Anatomical Therapeutic Class

bAb binding antibody BMI body mass index

BLOQ below the lower limit of quantification

CI confidence interval
COVID-19 coronavirus disease 2019
eCRF electronic case report form

eDiary electronic diary FAS full analysis set

GMFR geometric mean fold rise
GMT geometric mean titer

IM Intramuscular

IMP investigational medicinal product LLOQ lower limit of quantification

LOD limit of detection

MAAE medically-attended adverse event

MedDRA Medical Dictionary for Regulatory Activities

nAb neutralizing antibody
PPS per-protocol analysis set
PT Preferred Term (MedDRA)

S Spike

SAE serious adverse event

SARS-CoV-2 Severe Acute Respiratory Syndrome coronavirus-2

SAP statistical analysis plan
SCR seroconversion rate
SD standard deviation
SOC System Organ Class
ULN upper limit of normal
ULOQ upper limit of quantification
WHO World Health Organization

### 1.0 OBJECTIVES, ENDPOINTS AND ESTIMANDS

### 1.1 Objectives

### 1.1.1 Primary Objective

To evaluate the safety and immunogenicity of 2 doses of TAK-919 by intramuscular (IM) injection in healthy Japanese male and female adults aged  $\geq$  20 years, given 28 days apart.

### Safety:

To assess the safety of TAK-919 in terms of:

- Solicited local and systemic adverse events (AEs) for 7 days following each vaccination (day of vaccination + 6 subsequent days).
- Unsolicited AEs for 28 days following each vaccination (day of vaccination +27 subsequent days).
- Serious adverse events (SAEs), medically-attended adverse events (MAAEs), AEs leading to trial withdrawal or discontinuation of vaccination and Severe Acute Respiratory Syndrome coronavirus-2 (SARS-CoV-2) infection until Day 57.

### Immunogenicity:

To assess the immunogenicity of TAK-919 in terms of

• Serum binding antibody (bAb) levels against SARS-CoV-2 as measured by ligand-binding assay specific to the SARS-CoV-2 spike (S) protein on Day 57.

## 1.1.2 Secondary Objective(s)

### Safety:

To assess the safety of TAK-919 in terms of:

• SAEs, MAAEs, AEs leading to trial withdrawal or discontinuation of vaccination and SARS-CoV-2 infection throughout the trial.

### Immunogenicity:

To assess the immunogenicity of TAK-919 in terms of:

- Serum bAb levels against SARS-CoV-2 as measured by ligand-binding assay specific to the SARS-CoV-2 S protein on Day 29, Day 43, Day 209, and Day 394.
- Serum neutralizing antibody (nAb) titers against SARS-CoV-2 as measured by assay specific to wild-type virus on Day 29, Day 43, Day 57, Day 209, and Day 394.

## 1.1.3 Exploratory Objectives

### Immunogenicity:

To assess the immunogenicity of TAK-919 in terms of:

• Serum nAb levels against SARS-CoV-2 as measured by pseudovirus neutralization assays on Day 29, Day 43, Day 57, Day 209, and Day 394.

licable Terms of Use Post hoc exploratory immunogenicity data such as serum bAb levels against SARS-CoV-2 as measured by ligand-binding assay specific to the SARS-CoV-2 nucleocapsid protein may be generated using the residual of serum samples.

#### 1.2 **Endpoints**

#### 1.2.1 **Primary Endpoint(s)**

### Safetv:

- Percentage of subjects with reported solicited local AEs: injection site pain, erythema/redness, swelling, induration, and lymphadenopathy (axillary (underarm) swelling or tenderness ipsilateral to the side of injection) for 7 days following each vaccination (day of vaccination + 6 subsequent days).
- Percentage of subjects with solicited systemic AEs: headache, fatigue, myalgia, arthralgia, nausea/vomiting, chills, and fever for 7 days following each vaccination (day of vaccination + 6 subsequent days).
- Percentage of subjects with unsolicited AEs for 28 days after each vaccination.
- Percentage of subjects with SAE until Day 57.
- Percentage of subjects with MAAEs until Day 57.
- Percentage of subjects with any AE leading to discontinuation of vaccination.
- Percentage of subjects with any AE leading to subject's withdrawal from the trial until Day 57.
- Percentage of subjects with SARS-CoV-2 infection until Day 57.

## Immunogenicity:

Geometric mean titers (GMT), geometric mean fold rise (GMFR) and seroconversion rate (SCR; defined at percentage of subjects with a change from below the limit of detection (LOD) or the lower limit of quantification [LLOQ] to equal to or above LOD or LLOQ, OR,  $\geq 4$ -fold rises from baseline) of serum bAb against SARS-CoV-2 as measured by ligand-binding assay specific to the SARS-CoV-2 S protein on Day 57.

### Secondary Endpoint(s) 1.2.2

### Safety:

- Percentage of subjects with SAE throughout the trial.
- Percentage of subjects with MAAEs throughout the trial.
- Percentage of subjects with any AE leading to subject's withdrawal from the trial from the day of vaccination throughout the trial.
- Percentage of subjects with SARS-CoV-2 infection throughout the trial.

## Immunogenicity:

- GMT, GMFR and SCR of serum bAb against SARS-CoV-2 as measured by ligand-binding assay specific to the SARS-CoV-2 S protein on Day 29, Day 43, Day 209, and Day 394.
- AGMT, GMFR and SCR (defined at percentage of subjects with a change from below the LOD or LLOQ to equal & to or above LOD or LLOO, OR, ≥ 4-fold rises from baseline) of serum nAb against SARS-CoV-2 as measured by assay specific to wild-type virus on Day 29, Day 43, Day 57, Day 209, and Day 394.

#### 1.2.3 **Exploratory Endpoint(s)**

GMT, GMFR and SCR (defined at percentage of subjects with a change from below LOD or LLOO to equal to or above LOD or LLOO,  $OR \ge 4$ -fold rises from baseline) of serum nAb against SARS-CoV-2 as measured by pseudovirus neutralization assays on Day 29, Day 43, Day 57, Day 209, and Day 394.

reins of Use Additional immunogenicity data such as serum bAb levels against SARS-CoV-2 as measured by ligand-binding assay specific to the SARS-CoV-2 nucleocapsid protein may be evaluated using the residual of serum samples.

#### 2.0 STUDY DESIGN

This is a phase 1/2 randomized, observer-blind, placebo-controlled trial to evaluate the safety and immunogenicity of 2 doses of TAK-919 by IM injection in healthy Japanese male and female adults, given 28 days apart.

The trial is planned to enroll 200 subjects (150 subjects in the TAK-919 arm and 50 subjects in the placebo arm). Of them, 140 subjects will be stratified by age as  $\geq 20$  years to < 65 years (100) subjects in the TAK-919 arm and 40 subjects in the placebo arm), and 60 subjects will be stratified by age as  $\geq 65$  years (50 subjects in the TAK-919 arm and 10 subjects in the placebo arm).

Once all screening assessments following informed consent are completed and eligibility is confirmed, the subject will receive the first dose of TAK-919 or saline placebo by IM injection on Day 1, and receive the second dose of TAK-919 or saline placebo after 28 days of the first vaccination (Day 29). All subjects will be followed up for safety and immunogenicity for 12 months after the last trial vaccination.

Each subject will be provided with an electronic diary (eDiary). Oral body temperature, and solicited local and systemic AEs will be recorded in the eDiary by the subjects for 7 days after each vaccination (including the day of vaccination). All subjects will be followed for unsolicited AEs for 28 days following each vaccination (day of vaccination +27 subsequent days). All subjects will be followed for SAEs, MAAEs, and AEs leading to trial withdrawal or discontinuation of dosing during the trial. All subjects will also be tested for SARS-CoV-2 infection at prespecified time points (Day 1, Day 29, Day 57) and in case of suspected for COVID-19 clinical symptoms throughout the trial.

The primary analysis will be performed for safety and immunogenicity after all subjects have completed the Day 57 visit. After the primary analysis, the trial will be unblinded for Sponsor personnel. The Investigator, site staff and subjects will remain blinded to the investigational medicinal product (IMP) for 12 months after the last trial vaccination.

A schematic of the trial design is included as Figure 2.a.

Schedule of events can be found in protocol Section 2.1.

Figure 2.a Schematic of Trial Design



Abbreviations: COVID-19=coronavirus disease 2019, N/n=number of subjects.

### 3.0 STATISTICAL HYPOTHESES AND DECISION RULES

## 3.1 Statistical Hypotheses

Not Applicable.

### 3.2 Statistical Decision Rules

Not Applicable.

## 3.3 Multiplicity Adjustment

Given the exploratory nature of this study, no adjustment for multiple comparisons and multiplicity will be performed. That is, only nominal p-values will be provided if applicable.

No statistical testing will be performed for the safety endpoints.

### 4.0 SAMPLE-SIZE DETERMINATION

The objective of this trial is to evaluate the safety and immunogenicity of TAK-919 in the Japanese population. This trial is designed to be descriptive, and therefore the sample size was not determined based on formal statistical power calculations. The sample size for the trial is based on clinical and practical consideration and is considered sufficient to evaluate the objective of the trial. With 150 subjects in the TAK-919 group, the probability to observe at least one AE of 2% event rate is 95%. Considering the risk of disease burden of COVID-19, the number of placebo group in this trial was set as minimum as possible especially in the subjects  $\geq$  65 years old.

### 5.0 ANALYSIS SETS

The Full Analysis Set (FAS), Per-protocol Set (PPS) and Safety Analysis Set are defined for this trial. The FAS is defined as all randomized subjects who receive at least 1 dose of the treatment. Immunogenicity analyses will be conducted using the PPS defined to include subjects in the FAS and who have evaluable immunogenicity data and do not have significant protocol deviations which influence the immunogenicity assessment. Safety analyses will be conducted using the Safety Analysis Set defined as all subjects who receive at least 1 dose of the treatment.

Subject evaluability criteria for each analysis set will be fixed before unblinding of IMP assignment.

## 5.1 All Screened Subjects Analysis Set

The All Screened Subjects Analysis Set will consist of all subjects who provide informed consent for this study, to be used for reporting disposition and screening failures.

### 5.2 Safety Analysis Set

The Safety Analysis Set will consist of all subjects who receive at least 1 dose. Subjects will be analyzed according to the vaccine actually received. If 1st treatment is different from 2nd treatment due to error, subjects who receive at least one Active treatment is treated as "TAK-919".

### 5.3 Full Analysis Set

FAS will consist of all randomized subjects who receive at least 1 dose of the treatment. Subjects will be analyzed according to the study vaccine that the subject was randomized to receive and not according to what was actually received.

# 5.4 Per-Protocol Analysis Set

PPS will consist of all subjects who include in the FAS and who have evaluable immunogenicity data and do not have below significant protocol deviations which influence the immunogenicity assessment. Subjects with other protocol deviations might be excluded as necessary. Subjects will be analyzed according to the study vaccine that the subject was randomized to receive and not according to what was actually received.

- Missed dose of any planned injections
- Usage of prohibited medications specified in the protocol (section 7.3)
- Confirmation of SARS-CoV-2 infection before the 1<sup>st</sup> injection
- Out of allowance of blood sampling for immunogenicity on Day 57

General Considerations

Baseline values are defined as the last observed value before the first dose of study intervention.

Where applicable, variables will be summarized descriptively by study visit. For the variables, the counts and proportions of each possible value.

The denominator for the proportion is non-mission. non-missing responses to the categorical variable. For continuous variables, the number of subjects with non-missing values, mean, median, SD, minimum, and maximum values will be tabulated.

Study Day will be calculated from the reference start date and will be used to show start/stop day of assessments and events. Study day will be calculated relative to the first study intervention

• If assessment date is on or after the first study intervention date, then

Study Day = Assessment Date - First Study Intervention Date + 1

• Otherwise, Study Day = Assessment Date – First Study Intervention Date

In addition, day relative to vaccination will be derived for each vaccination dose. For example, day relative to the first dose will be equal to the Study Day. Day relative to the second dose will start with a value of 1 on the day of the second dose.

In the situation where the event date is partial or missing, Study Day and any corresponding durations will appear partial or missing in the listings.

For GMT, GMFR and SCR calculations, antibody values reported as below LLOQ will be replaced by  $0.5 \times LLOQ$  as applicable. Values that are greater than the upper limit of quantification (ULOQ) will be replaced by the ULOQ as applicable but will be listed as reported in the raw data. Same manner is applied for LOD. Values of blood sampling for immunogenicity after confirmation of SARS-CoV-2 infection will be excluded. Missing results will not be imputed. No other imputations will be performed.

A windowing convention will be used to determine the analysis value for a given study visit for immunogenicity analyses (Refer to Section 9.2.4).

Change from baseline will be calculated as:

Change from baseline = Test value at post-baseline visit – Baseline value

### **Handling of Treatment Misallocations**

All analyses using FAS and PPS will be performed as randomized, the other analysis will be performed as actually received, unless otherwise specified.

Number of subjects screened will be presented for the All Screened Subjects Analysis Set.

Number and percentages of subjects with screen failure and reason for screen failure will also be presented based on the All Screened Subjects Analysis Set. A listing will present subjects not meeting all eligibility criteria with the details of criteria not met.

Number of subjects are all subjects are all subjects and subjects are all s

Number of subjects randomized will be presented overall and by randomized group for the All Screened Subjects Analysis Set. Number of subjects randomized but not vaccinated will also be presented overall and by randomized group for the All Screened Subjects Analysis Set.

Number and percentages of subjects vaccinated will be presented overall and by treatment group for the Safety Analysis Set. Number and percentages of subjects who completed full course of study intervention, who discontinued early from study intervention (including reason for withdrawal), and who completed/discontinued early from the study (including reason for withdrawal) will be provided based on the Safety Analysis Set.

Similar summaries will be provided for each dose:

- Number and percentages of subjects vaccinated for first dose, ongoing in study after first dose, and discontinued early from the study (including reason for withdrawal) before second dose will be presented based on the Safety Analysis Set.
- Number and percentages of subjects vaccinated for second dose, ongoing in study (for primary analysis only) after second dose and discontinued early from the study (including reason for withdrawal) before 28 days post second dose and who discontinued early from the study (including reason for withdrawal) after 28 days (including 28 days) post second dose will be presented based on the Safety Analysis Set.

The analysis of number of ongoing subjects after first or second dose will only be presented for primary analysis and will not be included in the final analysis.

Number of subjects included and excluded from each analysis set (including reason for exclusion) will be summarized overall and by treatment group based on the All Screened Subjects Analysis Set. A listing showing inclusion and exclusion of each subject from each analysis set, including reason for exclusion, will be provided.

Number and percentage of subjects with important protocol deviations, as identified by the study team in a blinded manner as being major or critical, will be provided overall and by treatment group based on the Safety Analysis Set for each category specified in the Protocol Deviations Management Plan.

A listing of protocol deviations identified by the study team (important or not) will be provided.

# **Demographic and Other Baseline Characteristics**

### **Demographics**

Demographic data and other baseline characteristics will be presented for the Safety Analysis Set and PPS.

The following demographic and other baseline characteristics will be reported for this study:

- Age (years) at the date of signed informed consent
- Age group (years):  $20 \le 65$  and  $\ge 65$
- Age group (years):  $20 \le <65, 65 \le <75, 75 \le <85, \ge 85$
- Sex
- Race
- Weight (kg)
- Height (cm)
- Body mass index (BMI) (kg/m<sup>2</sup>)
- Seropositive status at baseline determined by serologic titer against SARS-CoV-2 nucleocapsid (Seronegative at baseline is defined as below limit of detection [LOD] or lower limit of quantification [LLOQ]) at Day 1. Seropositive at baseline is defined as equal to or above LOD or LLOQ at Day 1): Positive, Negative

Continuous demographic and other baseline characteristics will be summarised using descriptive statistics overall and by treatment group. Categorical demographic and other baseline characteristics using number and percentages of patients in each category overall and by treatment group. No statistical testing will be carried out for demographic or other baseline characteristics.

## 6.3.2 Medical History and Concurrent Medical Conditions

- Medical history is defined as any medical conditions/diseases that started and stopped prior to signing of informed consent.
- Concurrent medical conditions are defined as any medical conditions that started prior to signing of informed consent AND were ongoing at the time of signing of informed consent or ended on the day of signing of informed consent.

Medical history and concurrent medical conditions will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 23.0 or later, and will be summarized by System Organ Class (SOC) and Preferred Term (PT) based on the Safety Analysis Set. A subject having more than one medical condition within the same SOC/PT will be counted only once for that SOC or PT.

All medical history and concurrent medical conditions will be listed.

## 6.4 Medication History and Concomitant Medications

- Prior medications are defined as any medication that started and stopped prior to the first dose of study intervention.
- Concomitant medications are defined as:
  - Any medication that started before the first dose of study intervention AND was ongoing at the time of the first dose of study intervention;
  - Any medication that started on or after the day of first dose of study intervention.

Partially or completely missing medication start and stop dates will be handled as described in section 9.2.1.1.

All medications will be coded using the World Health Organization (WHO) Drug Global dictionary, version B3 March 2020 or later.


19-Mar-2021

Prior and concomitant medications will be summarized by Anatomical Therapeutic Class (ATC) level 2 and preferred drug name based on the Safety Analysis Set. A subject having more than one medication within the same ATC Level 2 or preferred drug name will be counted only once for that ATC Level 2 or preferred drug name.

All prior, concomitant medications and concomitant procedures will be listed.

6.5 Efficacy Analysis (Immunogenicity Analysis)

#### 6.5 **Efficacy Analysis (Immunogenicity Analysis)**

Unless otherwise specified, all summaries and figures for immunogenicity will be presented by treatment group, using the PPS and FAS.

#### 6.5.1 **Primary Endpoint(s) Analysis**

Geometric mean titers (GMT), geometric mean fold rise (GMFR) and seroconversion rate (SCR; defined at percentage of subjects with a change from below the limit of detection (LOD) or the limit of quantification (LLOO) to equal to or above LOD or LLOO. OR,  $\geq$  4-fold rises from baseline) of serum bAb against SARS-CoV-2 as measured by ligand-binding assay specific to the SARS-CoV-2 S protein on Day 57.

### Derivation of Endpoint(s) 6.5.1.1

Analyses will be conducted using the PPS and FAS.

SCR at Day 57 will be calculated along with its 95% confidence interval (CI) in each treatment group. For antibody titer values and the changes from baseline, GMT, GMFR, summary statistics and 95% CIs of each endpoint at Day 57 will be calculated in each treatment group.

### Main Analytical Approach 6.5.1.2

#### Seroconversion Rate 6.5.1.2.1

Seroconversion is a binary outcome where a success is when subjects with a change from below the LOD or LLOQ to equal to or above LOD or LLOQ, OR, ≥4-fold rises from baseline.

The number and proportion of subjects who have a seroconversion at Day 57 will be summarized for each treatment group. The summary will also include the 95% CI of the proportion of subjects achieving seroconversion at Day 57, calculated based on the Clopper-Pearson method. The number and percentage of subjects with fold-rise  $\geq 2$ , fold-rise  $\geq 3$ , and fold-rise  $\geq 4$  from baseline will be summarized with 95% CI calculated based on the Clopper-Pearson method.

#### 6.5.1.2.2 GMT and GMFR

GMT and GMFR will be calculated and will be summarized at Day 57.

Descriptive statistics for GMT and GMFR will include number of subjects, geometric mean, 95% CI, minimum and maximum and will be presented for each treatment group.

The GMT will be calculated as the anti-logarithm of  $\Sigma$  (common log transformed titer/n), i.e., as the anti-logarithm transformation of the mean of the log-transformed titer, where n is the number of participants with titer information.

The 95% CI will be calculated as the anti-logarithm transformation of the upper and lower limits for a two-sided CI for the mean of the log-transformed titers.

The fold rise is calculated as the ratio of the post-vaccination titer level to the pre-vaccination titer level. GMFR will be calculated as anti-logarithm of  $\Sigma$  (common log transformed (post-vaccination titer) pre-vaccination titer)/n). The 95% CIs for GMFR will be calculated similarly to those for GMT.

## 6.5.2 Secondary Endpoint(s) Analysis

- GMT, GMFR and SCR of serum bAb against SARS-CoV-2 as measured by ligand-binding assay specific to the SARS-CoV-2 S protein on Day 29, Day 43, Day 209, and Day 394.
- GMT, GMFR and SCR (defined at percentage of subjects with a change from below LLOQ to equal to or above LLOQ, OR, ≥ 4-fold rises from baseline) of serum nAb against SARS-CoV-2 as measured by assay specific to wild-type virus on Day 29, Day 43, Day 57, Day 209, and Day 394.

## 6.5.2.1 Derivation of Endpoint(s)

Analyses will be conducted using the PPS and FAS.

Seroconversion rate of each endpoint at each time point will be calculated along with its 95% CI in each treatment group. For antibody titer values and the changes from baseline, GMT, GMFR, summary statistics and 95% CIs of each endpoint at each time point will be calculated in each treatment group.

### 6.5.2.2 Main Analytical Approach

### 6.5.2.2.1 Seroconversion Rate

Seroconversion of serum bAb against SARS-CoV-2 as measured by ligand-binding assay specific to the SARS-CoV-2 S protein is defined in Section 6.5.1.2.1.

Seroconversion of serum nAb against SARS-CoV-2 as measured by assay specific to wild-type virus is defined is a binary outcome where a success is when subjects with a change from below LOD or LLOQ to equal to or above LOD or LLOQ, OR,  $\geq$  4-fold rises from baseline.

SCR of each endpoint at each time point will be performed the same analysis of the primary endpoint analysis, as Section 6.5.1.2.1. The number and percentage of subjects with fold-rise  $\geq$  2, fold-rise  $\geq$ 3, and fold- rise  $\geq$ 4 from baseline at Day 29 and Day 57 will be summarized with 95% CI calculated based on the Clopper-Pearson method.

### 6.5.2.2.2 GMTs and GMFRs

GMTs and GMFRs of each endpoint at each time point will be performed the same analysis of the primary endpoint analysis, as Section 6.5.1.2.2.

### 6.5.2.2.3 Mixed Model For Repeated Measures (MMRM)

The following analysis is performed only for bAb against SARS-CoV-2 as measured by ligand-binding assay specific to the SARS-CoV-2 S protein.

Mixed Effect Model for longitudinal data with fold increase from baseline in log transformed anti-body titers as dependent variable, and treatment groups, visit, treatment-by-visit, age group, and baseline log-transformed anti-body titers as independent variables and subject as a random effect. This analysis will be performed only when the proportion of subjects whose value of immunogenicity is LLOQ is less than 50% at any visit and any treatment group.

An unstructured covariance structure will be used to model the within-subject errors. A Kenward-Roger approximation will be used for the denominator degrees of freedom. If there is a convergence issue due to the unstructured covariance matrix, a compound symmetry covariance structure will be used to model the within-subject errors.

The geometric least squares mean (GLSM) and corresponding 2-sided 95% CI for the antibody titers for each treatment group will be provided by visit.

In addition, the ratio of GLSM and the corresponding 2-sided 95% CI will be provided to assess the treatment difference (TAK-919 vs. Placebo) at each visit. The GLSM, and corresponding 95% CI results in log transformed scale estimated from the model will be back transformed to obtain these estimates in the original scale. Geometric mean ratio (GMR), estimated by the ratio of GLSM and the corresponding 2 sided 95% CI will be provided to assess the treatment difference between TAK-919 group vs. placebo group at each visit.

# 6.5.3 Exploratory Endpoints Analysis

• GMT, GMFR and SCR (defined at percentage of subjects with a change from below LOD or LLOQ to equal to or above LOD or LLOQ, OR, ≥ 4-fold rises from baseline) of serum nAb against SARS-CoV-2 as measured by pseudovirus neutralization assays on Day 29, Day 43, Day 57, Day 209, and Day 394.

# 6.5.3.1 Derivation of Endpoint(s)

Analyses will be conducted using the PPS and FAS.

Seroconversion rate at each time point will be calculated along with its 95% CI in each treatment group. For antibody titer values and the changes from baseline, GMT, GMFR, summary statistics and 95% CIs of each endpoint at each time point will be calculated in each treatment group.

SCR at each time point will be performed the same analysis of the primary endpoint analysis, as Section 6.5.1.2.1.

6.5.3.2.2 GMTs and GMFRs

GMTs and GMTs

GMTs and GMFRs at each time point will be performed the same analysis of the primary endpoint analysis, as Section 6.5.1.2.2.

Assessment of the potential relationship between serum bAb antibody against SARS-6.5.3.3 CoV-2 and serum nAb antibody against SARS-CoV-2

> Spearman's rank correlation and Scatter plot for common log transformed serum bAb antibody titer and common log transformed serum nAb antibody titer will be provided using PPS by each Visit by Treatment group and age group.

#### 6.5.4 **Subgroup Analyses**

Perform subgroup analyses on the items described in Section 6.5.1, Section 6.5.2.2.1 and Section 6.5.2.2.2. Subgroup analyses will be conducted using the PPS.

The subgroup is:

- Age group (years): 20 < 65 and  $\ge 65$
- Sex: Male, Female
- Seropositive status at baseline determined by serologic titer against SARS-CoV-2 nucleocapsid (Seronegative at baseline is defined as below limit of detection [LOD] or lower limit of quantification [LLOQ]) at Day 1. Seropositive at baseline is defined as equal to or above LOD or LLOQ at Day 1): Positive, Negative

### Safety Analysis 6.6

All safety summaries will be presented by treatment group based on the Safety Analysis Set. There will be no statistical comparisons between the treatment groups for safety data.

The primary safety endpoints are:

- Percentage of subjects with reported solicited local AEs: injection site pain, erythema/redness, swelling, induration, and lymphadenopathy (axillary (underarm) swelling or tenderness ipsilateral to the side of injection) for 7 days following each vaccination (day of vaccination + 6 subsequent days).
- Percentage of subjects with solicited systemic AEs: headache, fatigue, myalgia, arthralgia, nausea/vomiting, chills and fever for 7 days following each vaccination (day of vaccination + 6 subsequent days).
- Percentage of subjects with unsolicited AEs for 28 days after each vaccination.
- Percentage of subjects with SAE until Day 57.
- Percentage of subjects with MAAEs until Day 57.
- Percentage of subjects with any AE leading to discontinuation of vaccination.
- Percentage of subjects with any AE leading to subject's withdrawal from the trial until Day 57.
- Percentage of subjects with SARS-CoV-2 infection until Day 57.

The secondary safety endpoints are:

- Percentage of subjects with MAAEs throughout the trial.

  Percentage of subjects with any AE leading to subject's withdrawal from the trial from the day of vaccination throughout the trial.

  Percentage of subjects with SARS-CoV-2 infection throughout the trial.

  Adverse Events

### 6.6.1

Unsolicited adverse events will be coded using the MedDRA dictionary, version 23.0 or later.

Only AEs that started or worsened in severity on or after the first dose of study intervention will be presented in the summary. A listing of all AEs including those prior to the first vaccination will be provided.

#### All Adverse Events 6.6.1.1

An overall summary of number and percentages of subjects within each of the categories described in the sub-sections below will be provided based on the Safety Analysis Set. Should a subject experience multiple events within a category, the subject will be counted only once for that category.

#### 6.6.1.1.1 Severity Grading for AEs

Severity is classed as mild/ moderate/ severe as defined in the protocol Section 10.2. AEs with a missing severity will be classified as severe. AEs will be collected on AE page of eCRF. Should a subject experience multiple events within a SOC or PT, only the subject's worst grade will be counted for that SOC or PT.

### AEs Related to Study Intervention 6.6.1.1.2

AEs related to study intervention, as indicated by the Investigator as "Causality" in eCRF, will be provided. AEs with a missing "Causality" will be classified as related.

Should a subject experience multiple events within a SOC or PT, only the subject's worst relationship will be counted for that SOC or PT.

## **Primary Safety Endpoints**

# Occurrence of Solicited AEs for 7 Days Following Each Vaccination

Subjects will record solicited local and systemic AEs (Table 6.a), and oral body temperature, for  $\overline{7}$  days following each vaccination (day of vaccination + 6 subsequent days) in the eDiary.

Severity grading of solicited AEs will occur automatically based on subject's entry into the eDiary according to the grading scales presented in Table 6.a modified from the Food and Drug Administration guidance (Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials)[1].

If a solicited local or systemic AE continues beyond 7 days after dosing, the subject will capture the AE in the eDiary until resolution. The solicited AEs recorded in eDiaries beyond Day 7 should be reviewed by the Investigator either via phone call or at the following trial visit.

Table 6.a Solicited Local (Injection Site) Reactions and Systemic AEs

| Local Reaction to Ir | ijectable Product | | | (0) |
|---|---|---|---|---|
| | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life-<br>threatening<br>(Grade 4) |
| Injection site pain | Does not interfere with activity | Repeated use of<br>nonnarcotic pain<br>reliever > 24 hours or<br>interferes with activity | Any use of narcotic pain reliever or prevents daily activity | Emergency room visit or hospitalization |
| Erythema/<br>redness <sup>a</sup> | 2.5 - 5 cm | 5.1 - 10 cm | > 10 cm | Necrosis or exfoliative dermatitis |
| Induration <sup>a</sup> | 2.5 - 5 cm | 5.1 - 10 cm | > 10 cm | Necrosis |
| Swelling <sup>a</sup> | 2.5 - 5 cm | 5.1 - 10 cm | > 10 cm | Necrosis |
| Lymphadenopathy<br>(Axillary swelling<br>or tenderness at the<br>same side of<br>injection site) | Does not interfere with activity | Repeated use of<br>nonnarcotic pain<br>reliever > 24 hours or<br>interferes with activity | Any use of narcotic pain reliever or prevents daily activity | Emergency room visit or hospitalization |
| Solicited Systemic A | <b>AEs</b> | 0 | | |
| Headache | No interference with activity | Repeated use of OTC<br>pain reliever > 24 hours<br>or some interference<br>with activity | Any use of prescription pain reliever or prevents daily activity | Emergency room visit or hospitalization |
| Fatigue | No interference with activity | Some interference with activity | Prevents daily activity | Emergency room visit or hospitalization |
| Myalgia | No interference with activity | Some interference with activity | Prevents daily activity | Emergency room visit or hospitalization |
| Arthralgia | No interference with activity | Some interference with activity | Prevents daily activity | Emergency room visit or hospitalization |
| Nausea/<br>vomiting | No interference with activity or 1-2 episodes/24 hours | Some interference with activity or > 2 episodes/24 hours | Prevents daily activity, requires outpatient intravenous hydration | Emergency room visit or<br>hospitalization for<br>hypotensive shock |
| Chills | No interference with activity | Some interference with activity, but no treatment required | Prevents daily activity or treatment required | Emergency room visit or hospitalization |
| Fever b | 38.0°C – 38.4°C | 38.5°C – 38.9°C | 39.0°C – 40.0°C | > 40.0°C |

Abbreviations: AE: adverse event, OTC: over-the-counter.

a In addition to grading the measure local reaction at the greatest single diameter, the measurement should be recorded as a continuous variable.

b Oral temperature; no recent hot or cold beverages.

They will not be assessed for relationship to study intervention because solicited AEs are expected to occur after vaccination.

Solicited AEs up to 7 days following each vaccination uses data collected by eDiary, on the other hands solicited AEs after 7 days following each vaccination uses data collected by eCRF.

Solicited AEs will be summarized for each day post-vaccination and the total duration (day of vaccination plus 6 subsequent days). For each interval, the count and percentages of subjects will be determined for each of the following categories: subjects evaluated, subjects without any events, subjects with any events, mild events, moderate events, severe events, and potentially life-threatening events. Subjects should not be double counted; therefore, the event of greatest severity will be used for subjects with more than 1 episode of the same event. Similar count and percentages of subjects will be presented for solicited local AEs and solicited systemic AEs.

Also Solicited AEs persisting beyond 7 days after vaccination will be summarized by severity for each vaccination. Subjects should not be double counted; therefore, the event of greatest severity will be used for subjects with more than 1 episode of the same event.

Quantitative and categorical summary of the day of first onset of each event and the number of days subjects reported experiencing each event will be presented. The number of days a subject reported experiencing an event is calculated as the total of all days the subject reported the event, regardless of whether the symptom was reported on consecutive days (e.g., a headache reported on Day 1, Day 3, and Day 4 would be included with a duration of 3 days).

A listing of all solicited AEs will be provided.

## 6.6.2.2 Occurrence of Unsolicited AEs for 28 Days After Each Vaccination

All AEs are considered to be unsolicited AEs unless categorized as solicited AEs recorded in an eDiary. All unsolicited AEs will be recorded from the start of each dose for 28 days post each dose of study intervention.

Number and percentages of subjects with at least one unsolicited AE will be presented by SOC and PT. Should a subject experience multiple events within a SOC or PT, the subject will be counted only once for that SOC or PT.

Number and percentage of subjects with at least one unsolicited AE will be presented by PT. Should a subject experience multiple events within a PT, the subject will be counted only once for that PT.

Number and percentage of subjects with at least one unsolicited AE will be broken down further by 28 days interval post each dose (based on the start date of the event), maximum severity (refer to Section 6.6.1.1.1), relationship to study intervention (refer to Section 6.6.1.1.2).

A listing of all unsolicited AEs will be provided.

### 6.6.2.3 Occurrence of Serious AEs Until Day 57

Serious adverse events are those events recorded as "Serious" on the AE page of the eCRF. Only SAEs that started or worsened in severity on or after the first dose of study intervention will be presented in the summary.

Should a subject experience multiple events within a SOC or PT, the subject will be counted only once for that SOC or PT. Number and percentage of subjects with at least one SAE will be broken down further by 28 days interval post each dose (based on the start date of the event).

A listing of all SAEs including those prior to the first vaccination will be provided.

## 6.6.2.4 Occurrence of Medically-Attended Adverse Events Until Day 57

MAAEs are defined as AEs leading to an unscheduled visit to or by a healthcare professional including visits to an emergency department, but not fulfilling seriousness criteria.

A summary of MAAEs by SOC and PT will be presented. Should a subject experience multiple events within a SOC or PT during an interval, the subject will be counted only once for that SOC or PT during that particular interval. The summary of MAAEs will be broken down further by 28 days interval post each dose (based on the start date of the event).

A listing of all MAAEs will be provided.

# 6.6.2.5 AEs Leading to Discontinuation of Vaccination

AEs leading to discontinuation of vaccination are recorded as "Drug Withdrawn" for the question "Action Taken with Study Treatment" on the AE pages of the eCRF. A summary of AEs leading to discontinuation of vaccination by SOC and PT will be presented. The summary of AEs leading to discontinuation of vaccination will be broken down further by 28 days interval post each dose (based on the start date of the event).

A listing of all AEs leading to discontinuation of vaccination will be provided.

## 6.6.2.6 AEs Leading to Subject's Withdrawal From the Trial Until Day 57

AEs leading to subject's withdrawal from the trial are recorded as "Yes" for the question "AE Caused Study Discontinuation?" on the AE pages of the eCRF. A summary of AEs leading to withdrawal from the trial by SOC and PT will be presented. The summary of AEs leading to subject's withdrawal from the trial will be broken down further by 28 days interval post each dose (based on the start date of the event).

A listing of all AEs leading to subject's withdrawal from the trial will be provided.

## 6.6.2.7 SARS-CoV-2 Infection Until Day 57.

The incidence of the first SARS-CoV-2 infection will be summarized by treatment group based on the Safety Analysis Set.

licable Terms of Use A subject who is found to be positive to COVID-19 based on the PCR testing of SARS-CoV-2 infection is considered as having SARS-CoV-2 infection.

A listing of the PCR testing of SARS-CoV-2 infection will be provided.

#### 6.6.3 Secondary safety endpoints

#### 6.6.3.1 Occurrence of Serious AEs Throughout the Trial

A summary of SAEs started on and after first dose of study intervention will be presented by SOC and PT throughout the trial. Should a subject experience multiple events within a SOC or PT, the subject will be counted only once for that SOC or PT.

A listing of all SAEs (including SAE started prior to the start of first dose of study intervention) will be provided.

This analysis will be conducted only at the Final analysis.

### Occurrence of MAAEs Throughout the Trial 6.6.3.2

A summary of MAAEs by SOC and PT throughout the trial will be presented. Should a subject experience multiple events within a SOC or PT, the subject will be counted only once for that SOC or PT.

A listing of all MAAEs will be provided.

This analysis will be conducted only at the Final analysis.

### AEs Leading to Subject's Withdrawal From the Trial From the Day of Vaccination 6.6.3.3 Throughout the Trial

AEs leading to subject's withdrawal from the trial are recorded as "Yes" for the question "AE Caused Study Discontinuation?" on the AE pages of the eCRF. A summary of AEs leading to withdrawal from the trial by SOC and PT will be presented.

A listing of all AEs leading to subject's withdrawal from the trial will be provided.

## This analysis will be conducted only at the Final analysis. SARS-CoV-2 Infection Throughout the Trial

The incidence of the first SARS-CoV-2 infection will be performed the same analysis of the primary safety analysis, as Section 6.6.2.7.

A subject who is found to be positive to COVID-19 based on the PCR testing of SARS-CoV-2 infection or seroconversion in serum bAb levels against SARS-CoV-2 as measured by ligandbinding assay specific to the SARS-CoV-2 nucleocapsid protein is considered as having SARS-CoV-2 infection.

Seroconversion in serum bAb levels against SARS-CoV-2 as measured by ligand-binding assay specific to the SARS-CoV-2 nucleocapsid protein is defined differently for participants who were seropositive or seronegative at baseline as below:

- Participants seronegative at Baseline (below limit of detection [LOD] or lower limit of quantification [LLOQ] in serum bAb levels against SARS-CoV-2 as measured by ligand-binding assay specific to the SARS-CoV-2 nucleocapsid protein): seropositive as measured by serum bAb levels against SARS-CoV-2 as measured by ligand-binding assay specific to the SARS-CoV-2 nucleocapsid protein on study
- Participants seropositive at Baseline: 4-fold or more increase in serum bAb levels against SARS-CoV-2 as measured by ligand-binding assay specific to the SARS-CoV-2 nucleocapsid protein

A listing of the PCR testing of SARS-CoV-2 infection and subjects who seroconversion subjects will be provided.

## 6.6.4 Other Adverse Event Safety Endpoint

## 6.6.4.1 Adverse Events with an Outcome of Death throughout the trial

AEs with an outcome of death are those events which are recorded as "Fatal" on the AE page of the eCRF.

A listing of all AEs with an outcome of death will be provided.

# 6.6.4.2 Unsolicited Adverse Events of Hypersensitivity

A summary of hypersensitivity AEs (refer to APPENDIX 9.2.6 for the list of SMQs) by PT throughout the trial will be presented. Should a subject experience multiple events within a PT, the subject will be counted only once for that PT.

A listing of all hypersensitivity AEs will be provided.

### 6.6.4.3 Related Unsolicited Adverse Events of Hypersensitivity

A summary of related hypersensitivity AEs by PT throughout the trial will be presented. Should a subject experience multiple events within a PT, the subject will be counted only once for that PT.

A listing of all related hypersensitivity AEs will be provided.

### 6.6.5 Other Safety Analysis

### 6.6.5.1 Laboratory Evaluations

Clinical chemistry and hematology will be performed as per the schedule of events (refer to protocol Section 2.1). Table 6.b lists the clinical safety laboratory tests that will be performed.

**Table 6.b Lists the Clinical Safety Laboratory Tests** 

| Hematology | Blood Chemistry | |
|---------------------------------|----------------------------------|-----|
| Hemoglobin, | Alanine aminotransferase (ALT) | |
| Hematocrit | Aspartate aminotransferase (AST) | |
| Platelet count | Alkaline phosphatase (ALP) | 70 |
| Complete white blood cell count | Total bilirubin | (0) |
| Prothrombin time | Urea (blood urea nitrogen) | 10 |
| Partial thromboplastin time | Creatinine | |
| _ | Lipase | |

Quantitative laboratory parameters reported as "< X", i.e., below the lower limit of quantification (BLOQ) or "> X", i.e., above the upper limit of quantification (ULOQ), will be converted to X for the purpose of quantitative summaries, but will be presented as recorded, i.e., as "< X" or "> X" in the listings.

The following summaries will be provided based on the Safety Analysis Set for each of blood chemistry and hematology laboratory parameter:

- Observed and change from baseline in Standard International (SI) units by visit;
- Categorical value according to FDA grading guidance (FDA 2007) toxicity grades (for quantitative parameters with available FDA toxicity grades; refer to APPENDIX 9.2.5) by visit;
- A listing of subjects with at least one observed value in alanine aminotransferase (ALT) value ≥ 3 x upper limit of normal (ULN) or aspartate aminotransferase (AST) value ≥ 3 x ULN together with total bilirubin value ≥ 2 x ULN will be provided.

Serology, pregnancy, and urine drug screen data will not be summarized

All laboratory data excluding urine drug screen data will be listed.

## 6.6.5.1.1 Laboratory Toxicity Grades

Quantitative laboratory parameters with available FDA toxicity grades will be categorized as follows where higher grades representing a more severe toxicity (refer to APPENDIX 9.2.5 for each parameter toxicity grade criteria). FDA grading will be categorized for laboratory parameters listed in Table 6.b:

- Grade 1 (i.e., mild);
- Grade 2 (i.e., moderate);
- Grade 3 (i.e., severe)
- Grade 4 (i.e., potentially life-threatening)

Although not defined in the FDA toxicity grading system, non-missing laboratory parameter results not meeting any of the 4 grades defined in the FDA toxicity grading system will be categorized as 'No Toxicity'.

## 6.6.5.2 Vital Sign Measurements

The following vital sign parameters will be collected for this study as per the schedule of events (refer to protocol Section 2.1):

- Systolic blood pressure (SBP) (mmHg)
- Diastolic blood pressure (DBP) (mmHg)
- Pulse rate (beats per minute [bpm])
- Body temperature (°C)
- Respiratory rate (beats per minute [bpm])

The following summaries will be provided based on the Safety Analysis Set for all scheduled visits.

- Observed and change from baseline by visit;
- Categorical value according to FDA grading guidance (FDA 2007) toxicity grades (for quantitative parameters with available FDA toxicity grades; refer to APPENDIX 9.2.5) by visit;

A listing of all vital sign data will also be provided.

### 6.6.5.2.1 Vital Sign Toxicity Grades

Vital sign toxicity grades will be performed the same analysis of laboratory toxicity grades, as Section 6.6.5.1.1. But Grade 4 is considered only for Fever due to the limited data collection.

## **6.6.6** Extent of Exposure and Compliance

### 6.6.6.1 Exposure to Study Intervention

Due to the simplicity of dosing for this study, exposure is summarized in the Disposition table. No other summary will be reported. A listing will provide exposure information for all subjects in the Safety Analysis Set.

Report of overdose and medication error, if any, will be listed for the Safety Analysis Set.

### 6.6.6.2 Compliance with Study Intervention

Compliance will not be calculated since subjects are vaccinated at most twice.

### 6.6.7 Subgroup Analyses

Perform subgroup analyses on the items described in Section 6.6.2.

The subgroup is:

- Age group (years):  $20 \le < 65$  and  $\ge 65$
- Sex: Male, Female
- Seropositive status at baseline determined by serologic titer against SARS-CoV-2 nucleocapsid (Seronegative at baseline is defined as below limit of detection [LOD] or lower limit of quantification [LLOQ]) at Day 1. Seropositive at baseline is defined as equal to or above LOD or LLOQ at Day 1): Positive, Negative

### 6.7 Interim Analyses

An interim analysis is not planned in the trial.

The primary analysis will be performed for safety and immunogenicity after all subjects have completed the Day 57 visit. After the primary analysis, the trial will be unblinded only for the

Sponsor personnel. The Investigator, site staff and subjects will remain blinded to the IMP until trial end (Day 394).

### 7.0 REFERENCES

1. Department of Health and Human Services (DHHS), Food and Drug Administration, Center for Biologics Evaluation and Research (US). Guidance for industry: Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials. September 2007 [cited 10 Apr 2020] [10 screens]. Available from: https://www.fda.gov/media/73679/download/BiologicsBloodVaccines/GuidanceCompliance RegulatoryInformation/Guidances/Vaccines/ucm091977.pdf

## 8.0 CHANGES TO PROTOCOL PLANNED ANALYSES

The definition of Seroconversion Rate for serum bAb against SARS-CoV-2 as measured by ligand-binding assay specific to the SARS-CoV-2 S protein

Before the change

Seroconversion of serum bAb against SARS-CoV-2 as measured by ligand-binding assay specific to the SARS-CoV-2 S protein is defined is a binary outcome where a success is when subjects with a change from below LOD to equal to or above LOD, OR,  $\geq$  4-fold rises from baseline.

After the change

Seroconversion of serum bAb against SARS-CoV-2 as measured by ligand-binding assay specific to the SARS-CoV-2 S protein is defined is a binary outcome where a success is when subjects with a change from below LOD or LLOQ to equal to or above LOD or LLOQ, OR,  $\geq$  4-fold rises from baseline.

Reason for the change

According to the immunogenicity data to be reported from serology laboratories, the definition of SCR was updated to 'the percentage of subjects with a change from below the limit of detection [LOD] or the lower limit of quantification [LLOQ] to equal to or above LOD or LLOQ, OR,  $\geq$  4-fold rises from baseline'

The definition of Seroconversion Rate for serum nAb against SARS-CoV-2 as measured by assay specific to wild-type virus

Before the change

Seroconversion of serum nAb against SARS-CoV-2 as measured by assay specific to wild-type virus is defined is a binary outcome where a success is when subjects with a change from below LLOQ to equal to or above LLOQ, OR,  $\geq$  4-fold rises from baseline.

After the change

Seroconversion of serum nAb against SARS-CoV-2 as measured by assay specific to wild-type virus is defined is a binary outcome where a success is when subjects with a change from below LOD or LLOQ to equal to or above LOD or LLOQ, OR,  $\geq 4$ -fold rises from baseline.

Reason for the change

According to the immunogenicity data to be reported from serology laboratories, the definition of SCR was updated to 'the percentage of subjects with a change from below the limit of detection [LOD] or the lower limit of quantification [LLOQ] to equal to or above LOD or LLOQ, OR, ≥ 4-fold rises from baseline'

#### 9.0 **APPENDIX**

### **Changes From the Previous Version of the SAP** 9.1 Not Applicable.

### 9.2 **Data Handling Conventions**

### 9.2.1

### 9.2.1.1

| - | or the lower lin | mit of quantification [LLOQ] to equal to or above LOD or a baseline' |
|---|---|---|
| <ul><li>9.0 APPEND</li><li>9.1 Change</li><li>Not Applicable.</li></ul> | | entions eting Conventions |
| 9.2.1 Gener | andling Conve<br>al Data Repor<br>al Date Conve | |
| Start Date | Stop Date | Action |
| | Known or ongoing | If medication stop date < study intervention start date, assign as prior; If medication start date < study intervention start date and (medication stop date ≥ study intervention start date or medication is ongoing at study intervention start date), assign as concomitant; If study intervention start date ≤ medication start date, assign as concomitant. |
| Known or before | Partial | If known components of medication stop date show that medication stopped before study intervention start date, assign as prior; If medication start date < study intervention start date and (known components of medication stop date show that medication stopped on or after study intervention start date), assign as concomitant; If study intervention start date ≤ medication start date, assign as concomitant. |

| Start Date | Stop Date | Action |
|---|---|---|
| | | If medication stop date is missing, then it can never be assigned as prior only; |
| | Missing, not ongoing | If medication start date < study intervention start date, assign as concomitant; |
| | | If study intervention start date ≤ medication start date, assign as concomitant. |
| | | If medication stop date < study intervention start date, assign as prior; |
| | Known or | If (known components of medication start date show that medication started before study intervention start date) and (medication stop date ≥ study |
| | ongoing | intervention start date or medication is ongoing at study intervention start date), assign as concomitant; |
| | | If known components of medication start date show that medication started on or after study intervention start date, assign as concomitant. |
| | | If known components of medication stop date show that medication stopped before study intervention start date, assign as prior; |
| Partial | Partial | If (known components of medication start date show that medication started before study intervention start date) and (known components of medication stop date show that medication stopped on or after study intervention start |
| | NON-COM | date), assign as concomitant; If known components of medication start date show that medication started on or after study intervention start date, assign as concomitant. |
| 6 | 5 | Cannot be assigned as prior only; |
| of akedai. | Missing, not ongoing | If known components of medication start date show that medication started before study intervention start date, assign as concomitant; |
| of St. | ongoing | If known components of medication start date show that medication started on or after study intervention start date, assign as concomitant. |
| Missing | Known or ongoing | If medication stop date < study intervention start date, assign as prior; If medication stop date >= study intervention start date or medication is ongoing at study intervention start date, assign as concomitant. |

| Start Date | Stop Date | Action |
|---|---|---|
| | Partial | If known components of medication stop date show that medication stopped before study intervention start date, assign as prior; If known components of medication stop date show that medication stopped on or after study intervention start date, assign as concomitant. |
| | Missing, not ongoing | Assign as concomitant. |

### 9.2.2 **Definition of Baseline**

Unless otherwise specified, baseline is defined as the last non-missing measurement taken prior to the first dose of study intervention (including unscheduled assessments). In the case where the last non-missing measurement and the date and time of the first dose of study intervention coincide, that measurement will be considered pre-baseline, but AEs and medications commencing on the date of the first dose of study intervention will be considered post-baseline.

## 9.2.3 Unscheduled Visits, and Early Termination Data

For by-visit summaries, data recorded at the nominal visit will be presented. That is, unscheduled, and early termination measurements will not be included in by-visit summaries but might contribute to the baseline timepoint and/or maximum value, where required (e.g. shift table). An exception to this rule applies to immunogenicity analysis as stated in Section 9.2.4.

Listings will include scheduled, unscheduled, retest and early discontinuation data.

### 9.2.4 Definition of Visit Windows

A windowing convention will be used to determine the analysis value for a given study visit for immunogenicity data analyses. The date will be used eCRF data.

The window conventions are:

- 1. A window of +/- 7 days from the target day is applied to the following visits: Study Days 29, 43, 57 (for Day 29, the date and time of second dose of study intervention can be used as upper bound);
- 2. A window of  $\pm$  30 days from the target day is applied to the following visits: Study Day 209 and Day 394;

Table 9.a Analysis Windows for Immunogenicity by Visit

| Dosing Period | Visit | Day Relative to Dose within the Dosing Period (b) | Visit Window (Study Day) Relative to the Dosing Period |
|---|---|---|---|
| Period 1 | Baseline (a) | ≤1 | ≤1 |
| (Relative to Dose 1) | Day 29 | 29 | 22 - 36 |
| Period 2 | Day 43 | 15 | 8 - 21 |
| (Relative to Dose 2) | Day 57 | 29 | 22 - 105 |
| | Day 209 | 181 | 106 - 273 |
| | Day 394 | 366 | 274 - 380 |

<sup>(</sup>a) Where time is available, the time of the collection must be prior to the first dose of study intervention. Day 1 observations taken after the first dose are considered post-baseline values.

One or more results for a particular immunogenicity variable may be obtained in the same visit window. In such an event, the result with the date closest to the expected visit date will be used in the analysis. In the event that two observations are equidistant from the expected visit date, the later observation will be used in the analysis.

Beside the immunogenicity analyses, no visit windowing will be performed for analysis of other variables in this study.

## 9.2.5 Tables for Laboratory and Vital Sign Abnormalities

The laboratory and vital sign values provided in the tables below serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate. For Vital Sign grading, Grade 4 is considered only for Fever due to the limited data collection.

<sup>(</sup>b) For each dosing period, the administration of the study intervention is designated as Study Day 1. For analyses within a period, the study day value is incremented by 1 for each date following the vaccine administration.

| 019 <i>–1501</i> | | | | |
|---|---|---|---|---|
| tical Analysis Plan 1.0 | | | | 19-Mar-2021 |
| | | | | Potentially Life |
| Vital Signs * | Mild (Grade 1) | Moderate(Grade 2) | Severe (Grade 3) | Potentially Life Threatening (Grade 4) |
| Fever (°C) **<br>(°F) ** | 38.0 - 38.4<br>100.4 - 101.1 | 38.5 - 38.9<br>101.2 - 102.0 | 39.0 - 40<br>102.1 - 104 | > 40<br>> 104 |
| Tachycardia - beats per<br>minute | 101 – 115 | 116 – 130 | > 130 | ER visit or<br>hospitalization for<br>arrhythmia |
| Bradycardia - beats per<br>minute*** | 50 – 54 | 45 – 49 | < 45 | ER visit or<br>hospitalization for<br>arthythmia |
| Hypertension (systolic) -<br>mm Hg | 141 – 150 | 151 – 155 | >155 | ER visit or hospitalization for malignant hypertension |
| Hypertension (diastolic) -<br>mm Hg | 91 – 95 | 96 – 100 | > 100 | ER visit or<br>hospitalization for<br>malignant<br>hypertension |
| Hypotension (systolic) –<br>mm Hg | 85 – 89 | 80 – 84 | € 80 | ER visit or<br>hospitalization for<br>hypotensive shock |
| Respiratory Rate - breaths<br>per minute | 17 – 20 | 21 – 25 | > 25 | Intubation |

Subject should be at rest for all vital sign measurements.

<sup>\*\*</sup> Oral temperature; no recent hot or cold beverages or smoking.

Ad to 1 . Ay subject p. Ay sub \*\*\* When resting heart rate is between 60 - 100 bears per minute. Use clinical judgement when characterizing bradycardia among some healthy subject populations, for example, conditioned athletes.

| Serum * | Mild (Grade 1) | Moderate | Severe | Potentially Life |
|---|---|---|---|---|
| | | (Grade 2) | (Grade 3) | Threatening<br>(Grade 4)** |
| Sodium - Hyponatremia mEq/L | 132 - 134 | 130 - 131 | 125 - 129 | < 125 |
| Sodium – Hypernatremia mEq/L | 144 – 145 | 146 – 147 | 148 - 150 | > 150 |
| Potassium – Hyperkalemia mEq/L | 5.1 – 5.2 | 5.3 - 5.4 | 5.5 - 5.6 | > 5.6 |
| Potassium – Hypokalemia mEq/L | 3.5 – 3.6 | 3.3 – 3.4 | 3.1 – 3.2 | < 3.1 |
| Glucose – Hypoglycemia mg/dL | 65 – 69 | 55 – 64 | 45 – 54 | < 45 |
| Glucose – Hyperglycemia | | | | Insulin |
| Fasting – mg/dL | 100 - 110 | 111 – 125 | >125 | requirements or |
| Random – mg/dL | 110 – 125 | 126 – 200 | >200 | hyperosmolar<br>coma |
| Blood Urea Nitrogen<br>BUN mg/dL | 23 – 26 | 27 – 31 | > 31 | Requires<br>dialysis |
| Creatinine – mg/dL | 1.5 – 1.7 | 1.8 - 2.0 | 2.1 – 2.5 | > 2.5 or requires<br>dialysis |
| Calainm himagalaamia ma/dI | 8.0 - 8.4 | 7.5 – 7.9 | 7.0 = 7.4 | < 7.0 |
| Calcium - hypocalcemia mg/dL | | | 14.6 - 12.0 | |
| Calcium - hypercalcemia mg/dL | 10.5 - 11.0 | 11.1 - 11.5 | 0.9 – 1.0 | > 12.0 |
| Magnesium – hypomagnesemia mg/dL<br>Phosphorous – hypophosphatemia<br>mg/dL | 1.3 – 1.5<br>2.3 – 2.5 | 1.1 – 1.2<br>2.0 – 2.2 | 1.6 – 1.9 | < 0.9<br>< 1.6 |
| CPK – mg/dL | 1.25 – 1.5 x<br>ULN*** | 1.6 - 3.0 x ULN | 3.1 –10 x ULN | > 10 x ULN |
| Albumin - Hypoalbuminemia g/dL | 2.8 - 3.1 | 2.5 - 2.9 | < 2.5 | |
| Total Protein - Hypoproteinemia g/dL | 5.5 - 6.0 | 5.0-5.4 | < 5.0 | |
| Alkaline phosphate –<br>increase by factor | 1.1 – 2.0 x ULN | 3.0 x ULN | .3.1-10 x ULN | > 10 x ULN |
| Liver Function Tests -ALT, AST increase by factor | 1.1 – 2.5 x UIA | 2.6 - 5.0 x ULN | 5.1 – 10 x ULN | > 10 x ULN |
| Bilirubin - when accompanied | 1.1 - 1.25 x ULN | 1.26 - 1.5 x ULN | 1.51 - 1.75 x ULN | > 1.75 x ULN |
| by any increase in Liver Function Test<br>increase by factor | | | | |
| Bilirubin – when Liver Function Test<br>is normal; increase by factor | 1.5 x ULN | 1.6 – 2.0 x ULN | 2.0 - 3.0 x ULN | > 3.0 x ULN |
| Cholesterol | 201 – 210 | 211 – 225 | > 226 | |
| Pancreatic enzymes - amylase, lipase | 1.1 – 1.5 x ULN | 1.6 - 2.0 x ULN | 2.1 – 5.0 x ULN | > 5.0 x ULN |
| parameters. Institutional normal refe ** The clinical signs or symptoms asso laboratory abnormalities as Potential within a grade 3 parameter (125-129 new seizure associated with the low ***ULN" is the upper limit of the norm | ciated with laboratory<br>lly Life Threatening (<br>mE/L) should be reco<br>sodium value. | abnormalities might<br>Grade 4). For examp | result in characterizati<br>le. a low sodium value | ion of the<br>that falls |

<sup>\*</sup> The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate.

<sup>\*\*</sup> The clinical signs or symptoms associated with laboratory abnormalities might result in characterization of the laboratory abnormalities as Potentially Life Threatening (Grade 4). For example, a low sodium value that falls within a grade 3 parameter (125-129 mE/L) should be recorded as a grade 4 hyponatremia event if the subject had a

| Hematology * | Mild (Grade 1) | Moderate<br>(Grade 2) | Severe (Grade 3) | Potentially Life<br>Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Hemoglobin (Female) - gm/dL | 11.0 - 12.0 | 9.5 - 10.9 | 8.0 - 9.4 | < 8.0 |
| Hemoglobin (Female) | Any decrease - 1.5 | 1.6 - 2.0 | 2.1 - 5.0 | > 5.0 |
| change from baseline value - gm/dL | | | | |
| Hemoglobin (Male) - gm/dL | 12.5 - 13.5 | 10.5 - 12.4 | 8.5 - 10.4 | < 8.5 |
| Hemoglobin (Male) | Any decrease - 1.5 | 1.6 - 2.0 | 2.1 - 5.0 | > 5.0 |
| change from baseline value - gm/dL | | | | 60. |
| WBC Increase - cell/mm <sup>3</sup> | 10,800 - 15,000 | 15,001 - 20,000 | 20,001 - 25,000 | > 25,000 |
| WBC Decrease - cell/mm <sup>3</sup> | 2,500 - 3,500 | 1,500 - 2,499 | 1,000 - 1,499 | < 1,000 |
| Lymphocytes Decrease - cell/mm <sup>3</sup> | 750 - 1,000 | 500 - 749 | 250 - 499 | < 250 |
| Neutrophils Decrease - cell/mm3 | 1,500 - 2,000 | 1,000 - 1,499 | 500 – 999 | Q 500 |
| Eosinophils - cell/mm <sup>3</sup> | 650 - 1500 | 1501 - 5000 | > 5000 | Hypereosinophilic |
| Platelets Decreased - cell/mm <sup>3</sup> | 125,000 - 140,000 | 100,000 - 124,000 | 25,000 - 99,000 | < 25,000 |
| PT - increase by factor | 1.0 - 1.10 x | 1.11 - 1.20 x ULN | 1.21 - 1.21 DULN | > 1.25 ULN |
| (prothrombin time) | ULN** | | X V | |
| PTT - increase by factor | 1.0 - 1.2 x ULN | 1.21 - 1.4 x ULN | 1.41 - 1.5 x ULN | > 1.5 x ULN |
| (partial thromboplastin time) | | | .0 | |
| Fibrinogen increase - mg/dL | 400 - 500 | 501 – 600 | ≥600 | |
| Fibrinogen decrease - mg/dL | 150 - 200 | 125 - 149 | 100 – 124 | < 100 or associated |
| | | 125-149 | | with gross bleeding |
| | | .~0. | | or disseminated |
| | | | | intravascular |
| | | \ | | coagulation (DIC) |

The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate. "ULN" is the upper limit of the normal range.

### 9.2.6 Tables for Unsolicited Adverse Events of Hypersensitivity

Hypersensitivity are defined by the narrow terms pertaining to hypersensitivity SMQs in the tables below for a full list of preferred terms.

| PT Code | PT Term(English) |
|----------|--------------------------------------------|
| 10081035 | Acquired C1 inhibitor deficiency |
| 10048799 | Acute generalised exanthematous pustulosis |
| 10069773 | Administration related reaction |
| 10075096 | Administration site dermatitis |
| 10075099 | Administration site eczema |
| 10075102 | Administration site hypersensitivity |
| 10071156 | Administration site rash |
| 10075964 | Administration site recall reaction |
| 10075109 | Administration site urticaria |
| 10075969 | Administration site vasculitis |
| 10052613 | Allergic bronchitis |

| <i>TAK-919–1</i><br>Statistical <i>I</i> | <i>501</i><br>Analysis Plan 1.0 | 19-Mar-2021 Terms of Use applicable appl | C: |
|---|---|---|---|
| PT Code | PT Term(English) | . 5 | 2 |
| 10059447 | Allergic colitis | Ŏ. | |
| 10053779 | Allergic cough | "Us | |
| 10051394 | Allergic cystitis | <b>₹</b> ◎` | |
| 10075185 | Allergic eosinophilia | 2/6 | |
| 10075308 | Allergic gastroenteritis | ico. | |
| 10071198 | Allergic hepatitis | OPI | |
| 10057380 | Allergic keratitis | (O) | |
| 10060934 | Allergic oedema | "KL" | |
| 10075072 | Allergic otitis externa | | |
| 10061557 | Allergic otitis media | Sie | |
| 10050639 | Allergic pharyngitis | | |
| 10078853 | Allergic reaction to excipient Allergic respiratory disease | | |
| 10063532 | Allergic respiratory disease | | |
| 10063527 | Allergic respiratory symptom | | |
| 10049153 | Allergic sinusitis | | |
| 10079554 | Allergic stomatitis | | |
| 10066173 | Allergic transfusion reaction | | |
| 10075479 | Allergy alert test positive | | |
| 10056352 | Allergy test positive | | |
| 10074079 | Allergy to immunoglobulin therapy | | |
| 10077279 | Allergy to surgical sutures | | |
| 10055048 | Allergy to vaccine | | |
| 10078682 | Anal eczema | | |
| 10002198 | Anaphylactic reaction | | |
| 10002199 | Anaphylactic shock | | |
| 10067113 | Anaphylactic transfusion reaction | | |
| 10002216 | Anaphylactoid reaction | | |
| 10063119 | Anaphylactoid shock | | |
| 10002222 | Anaphylaxis treatment | | |
| 10002424 | Angioedema | | |
| | 1 | | |

| | • |
|----------|----------------------------------------------------------|
| PT Code | PT Term(English) |
| 10064059 | Antiallergic therapy |
| 10065514 | Antiendomysial antibody positive |
| 10050894 | Anti-neutrophil cytoplasmic antibody positive vasculitis |
| 10003036 | Application site dermatitis |
| 10050099 | Application site eczema |
| 10063683 | Application site hypersensitivity |
| 10003054 | Application site rash |
| 10076024 | Application site recall reaction |
| 10050104 | Application site urticaria |
| 10076027 | Application site vasculitis |
| 10061430 | Arthritis allergic |
| 10075084 | Aspirin-exacerbated respiratory disease |
| 10081492 | Atopic cough |
| 10003645 | Atopy |
| 10005149 | Blepharitis allergic |
| 10005589 | Blood immunoglobulin E abnormal |
| 10005591 | Blood immunoglobulin E increased |
| 10006404 | Bromoderma |
| 10006482 | Bronchospasm |
| 10083809 | Bullous haemorrhagic dermatosis |
| 10073992 | Catheter site dermatitis |
| 10073995 | Catheter site eczema |
| 10073998 | Catheter site hypersensitivity |
| 10052271 | Catheter site rash |
| 10052272 | Catheter site urticaria |
| 0074014 | Catheter site vasculitis |
| 10071399 | Chronic eosinophilic rhinosinusitis |
| 10071380 | Chronic hyperplastic eosinophilic sinusitis |
| 10009192 | Circulatory collapse |
| 10052250 | Circumoral oedema |

Whiled to the applicable Terms of Use

| TAK-919-1<br>Statistical A | <i>501</i><br>Analysis Plan 1.0 | 19-Mar-2021 Joje Ct. to the applicable |
|---|---|---|
| PT Code | PT Term(English) | |
| 10081703 | Circumoral swelling | |
| 10010726 | Conjunctival oedema | |
| 10010744 | Conjunctivitis allergic | <∞, |
| 10067510 | Contact stomatitis | % |
| 10066973 | Contrast media allergy | iicat |
| 10010836 | Contrast media reaction | ·06// |
| 10011033 | Corneal oedema | O. O. |
| 10011686 | Cutaneous vasculitis | FIL. |
| 10062918 | Dennie-Morgan fold | <i>A</i> . 10 |
| 10012431 | Dermatitis | Nie V |
| 10012432 | Dermatitis acneiform | 77' |
| 10012434 | Dermatitis allergic | |
| 10012438 | Dermatitis atopic | |
| 10012441 | Dermatitis bullous | |
| 10012442 | Dermatitis contact | |
| 10012455 | Dermatitis exfoliative | |
| 10012456 | Dermatitis exfoliative generalised | |
| 10012468 | Dermatitis herpetiformis | |
| 10012470 | Dermatitis infected | |
| 10058675 | Dermatitis psoriasiform | |
| 10072867 | Device allergy | |
| 10076665 | Dialysis membrane reaction | |
| 10070559 | Distributive shock | |
| 10076470 | Documented hypersensitivity to administered product | |
| 10013687 | Drug eruption | |
| 10013700 | Drug hypersensitivity | |
| 10074350 | Drug provocation test | |
| 10073508 | Drug reaction with eosinophilia and systemic symptoms | |
| 10014184 | Eczema | |
| 10014198 | Eczema infantile | |

| | • |
|----------|-----------------------------------------------|
| PT Code | PT Term(English) |
| 10014201 | Eczema nummular |
| 10066042 | Eczema vaccinatum |
| 10058681 | Eczema vesicular |
| 10055182 | Eczema weeping |
| 10056387 | Encephalitis allergic |
| 10014627 | Encephalopathy allergic |
| 10078117 | Eosinophilic granulomatosis with polyangiitis |
| 10059284 | Epidermal necrosis |
| 10053177 | Epidermolysis |
| 10014989 | Epidermolysis bullosa |
| 10015029 | Epiglottic oedema |
| 10015218 | Erythema multiforme |
| 10015226 | Erythema nodosum |
| 10064579 | Exfoliative rash |
| 10015907 | Eye allergy |
| 10052139 | Eye oedema |
| 10015967 | Eye swelling |
| 10015993 | Eyelid oedema |
| 10016029 | Face oedema |
| 10016741 | Fixed eruption |
| 10018258 | Giant papillary conjunctivitis |
| 10049305 | Gingival oedema |
| 10018291 | Gingival swelling |
| 10066837 | Gleich's syndrome |
| 10059499 | Haemorrhagic urticaria |
| 10058898 | Hand dermatitis |
| 10019617 | Henoch-Schonlein purpura |
| 10069440 | Henoch-Schonlein purpura nephritis |
| 10062506 | Heparin-induced thrombocytopenia |
| 10019860 | Hereditary angioedema |

Whiled to the applicable Terms of Use

| | • | |
|----------|-------------------------------------------------------------|----|
| PT Code | PT Term(English) | |
| 10080955 | Hereditary angioedema with C1 esterase inhibitor deficiency | |
| 10020751 | Hypersensitivity | |
| 10081004 | Hypersensitivity myocarditis | |
| 10081988 | Hypersensitivity pneumonitis | |
| 10020764 | Hypersensitivity vasculitis | |
| 10021247 | Idiopathic urticaria | |
| 10067142 | Immediate post-injection reaction | |
| 10083842 | Immune thrombocytopenia | |
| 10070581 | Immune tolerance induction | |
| 10063855 | Implant site dermatitis | 11 |
| 10063858 | Implant site hypersensitivity | |
| 10063786 | Implant site rash | |
| 10063787 | Implant site urticaria | |
| 10073168 | Incision site dermatitis | |
| 10073411 | Incision site rash | |
| 10082742 | Infusion related hypersensitivity reaction | |
| 10051792 | Infusion related reaction | |
| 10065458 | Infusion site dermatitis | |
| 10074850 | Infusion site eczema | |
| 10065471 | Infusion site hypersensitivity | |
| 10059830 | Infusion site rash | |
| 10076085 | Infusion site recall reaction | |
| 10065490 | Infusion site urticaria | |
| 10074851 | Infusion site vasculitis | |
| 10071152 | Injection related reaction | |
| 10022056 | Injection site dermatitis | |
| 10066221 | Injection site eczema | |
| 10022071 | Injection site hypersensitivity | |
| 10022094 | Injection site rash | |
| | 1 | ı |

This of Use applicable Terms of Use

| | • |
|----------|---------------------------------------|
| PT Code | PT Term(English) |
| 10066797 | Injection site recall reaction |
| 10022107 | Injection site urticaria |
| 10067995 | Injection site vasculitis |
| 10073612 | Instillation site hypersensitivity |
| 10073622 | Instillation site rash |
| 10073627 | Instillation site urticaria |
| 10067972 | Interstitial granulomatous dermatitis |
| 10076229 | Intestinal angioedema |
| 10052098 | Iodine allergy |
| 10051891 | Kaposi's varicelliform eruption |
| 10069167 | Kounis syndrome |
| 10023845 | Laryngeal oedema |
| 10064866 | Laryngitis allergic |
| 10023891 | Laryngospasm |
| 10023893 | Laryngotracheal oedema |
| 10070492 | Limbal swelling |
| 10024558 | Lip oedema |
| 10024570 | Lip swelling |
| 10076606 | Mast cell degranulation present |
| 10075572 | Medical device site dermatitis |
| 10075575 | Medical device site eczema |
| 10075579 | Medical device site hypersensitivity |
| 10075585 | Medical device site rash |
| 10076140 | Medical device site recall reaction |
| 10075588 | Medical device site urticaria |
| 10075203 | Mouth swelling |
| 10056671 | Mucocutaneous rash |
| 10028164 | Multiple allergies |
| 10029120 | Nephritis allergic |
| 10029415 | Nikolsky's sign |

Juliect to the applicable Terms of Use

| statistical 1 | 111a1y 515 1 1a11 1.0 |
|---------------|-------------------------------------------------|
| PT Code | PT Term(English) |
| 10075807 | Nodular rash |
| 10084049 | Nutritional supplement allergy |
| 10030081 | Oculomucocutaneous syndrome |
| 10067317 | Oculorespiratory syndrome |
| 10030110 | Oedema mouth |
| 10068355 | Oral allergy syndrome |
| 10067950 | Oropharyngeal blistering |
| 10078783 | Oropharyngeal oedema |
| 10031111 | Oropharyngeal spasm |
| 10031118 | Oropharyngeal swelling |
| 10056998 | Palatal oedema |
| 10074403 | Palatal swelling |
| 10068809 | Palisaded neutrophilic granulomatous dermatitis |
| 10056872 | Palpable purpura |
| 10074332 | Pathergy reaction |
| 10034541 | Perioral dermatitis |
| 10034545 | Periorbital oedema |
| 10056647 | Periorbital swelling |
| 10034829 | Pharyngeal oedema |
| 10082270 | Pharyngeal swelling |
| 10080894 | Procedural shock |
| 10063438 | Pruritus allergic |
| 10037789 | Radioallergosorbent test positive |
| 10037844 | Rash |
| 10037855 | Rash erythematous |
| 10037857 | Rash follicular |
| 10037867 | Rash macular |
| 10037868 | Rash maculo-papular |
| 10050004 | Rash maculovesicular |
| 10037870 | Rash morbilliform |

Whiled to the applicable Terms of Use

| <i>TAK-919–1</i><br>Statistical <i>A</i> | <i>501</i><br>Analysis Plan 1.0 | 19-Mar-2021 Of Use applicable to the applicable to |
|---|---|---|
| | I man and the | 150 |
| PT Code | PT Term(English) | |
| 10037871 | Rash neonatal | |
| 10037879 | Rash papulosquamous | SIM |
| 10037884 | Rash pruritic | 70 |
| 10037888 | Rash pustular | 2016 |
| 10057984 | Rash rubelliform | i Car |
| 10037890 | Rash scarlatiniform | 08 |
| 10037898 | Rash vesicular | |
| 10037973 | Reaction to azo-dyes | in |
| 10037974 | Reaction to colouring | |
| 10079925 | Reaction to excipient | ie |
| 10037977 | Reaction to food additive | 26, |
| 10064788 | Reaction to preservatives Red man syndrome | |
| 10038192 | Red man syndrome | |
| 10039085 | Rhinitis allergic | |
| 10057431 | Scleral oedema | |
| 10051126 | Scleritis allergic | |
| 10083260 | Scrotal dermatitis | |
| 10039755 | Scrotal oedema | |
| 10040400 | Serum sickness | |
| 10040402 | Serum sickness-like feaction | |
| 10040560 | Shock | |
| 10040581 | Shock symptom | |
| 10083164 | SIS-TEN overlap | |
| 10040893 | Skin necrosis | |
| 10040914 | Skin reaction | |
| 10040934 | Skin test positive | |
| 10041307 | Solar urticaria | |
| 10041316 | Solvent sensitivity | |
| 10042033 | Stevens-Johnson syndrome | |
| 10074509 | Stoma site hypersensitivity | |
| 100/4507 | Sterm site hypersonautrity | |

| <i>TAK-919–1</i><br>Statistical <i>A</i> | <i>501</i><br>Analysis Plan 1.0 | 19-Mar-2021 Terrins of Use Applicable Applicable Joine applicable |
|---|---|---|
| PT Code | PT Term(English) | 1/56 |
| 10059071 | Stoma site rash | |
| 10042682 | Swelling face | 25 |
| 10042690 | Swelling of eyelid | * Off |
| 10042727 | Swollen tongue | \ <b>©</b> |
| 10078325 | Symmetrical drug-related intertriginous and flexural exanthema | ador |
| 10079645 | Therapeutic product cross-reactivity | |
| 10079043 | Tongue oedema | 200 |
| 10043967 | Toxic epidermal necrolysis | |
| | Toxic epidermai necrolysis | *0 |
| 10057970 | Toxic skin eruption | |
| 10044296 | Tracheal oedema | |
| 10045240 | Type I hypersensitivity | |
| 10054000 | | |
| 10053614 | | |
| 10053613 | Type IV hypersensitivity reaction | |
| 10046735 | Urticaria | |
| 10046740 | Urticaria cholinergic | |
| 10052568 | Urticaria chronic | |
| 10046742 | Urticaria contact | |
| 10046750 | Urticaria papular | |
| 10046751 | Urticaria physical | |
| 10046752 | Urticaria pigmentosa | |
| 10046755 | Urticaria vesiculosa | |
| 10082290 | Urticarial dermatitis | |
| 10048820 | Urticarial vasculitis | |
| 10069477 | Vaccination site dermatitis | |
| 10076161 | Vaccination site eczema | |
| 10069489 | Vaccination site exfoliation | |
| 10068880 | Vaccination site hypersensitivity | |
| 10069482 | Vaccination site rash | |
| 10076188 | Vaccination site recall reaction | |

| TAK-919-1<br>Statistical | 1501<br>Analysis Plan 1.0 | 19-Mar-2021 The applicable reins of Use |
|---|---|---|
| PT Code | PT Term(English) | , 1/9 |
| 10069622 | Vaccination site urticaria | 60 |
| 10076191 | Vaccination site vasculitis | in |
| 10069623 | Vaccination site vesicles | <∞, |
| 10046943 | Vaginal ulceration | 2/0 |
| 10047111 | Vasculitic rash | ;;c81 |
| 10081000 | Vernal keratoconjunctivitis | 00/1 |
| 10077117 | Vessel puncture site rash | |
| 10077813 | Vessel puncture site vesicles | |
| 10066273 | Vulval eczema | |
| 10047768 | Vulval ulceration | sie |
| 10071588 | Vulvovaginal rash | n, |
| 10050181 | Vulvovaginal ulceration | |
| 10080783 | Vulvovaginitis allergic | |

### **Programming Conventions for Output** 9.3

## **Dates & Times**

Depending on data available, dates and times will take the form yyyy-mm-dd hh:mm:ss.

### **Spelling Format**

English US.

## Paper size, Orientation, and Margins

The size of paper will be A4 and the page orientation will be landscape. Margins will provide at least 1 inch (2.54 centimeters) of white space all around the page.

### **Fonts**

The font type 'Courier New' will be used, with a font size of 8. The font color will be black with no bolding, underlining, italics or subscripting.

## **Presentation of Treatment Groups**

For outputs, treatment groups will be represented as follows and in the given order:

| Treatment Group | Tables and Graphs | Listings | |
|----------------------------|-------------------|----------|-----------------|
| Placebo | 1 | 1 | |
| TAK-919 | 2 | 2 | 44 |
| Randomized, Not Vaccinated | N/A | 3 | \ <sub>\O</sub> |
| Screen Failure | N/A | 4 | Ne |

## **Presentation of Nominal visits**

For outputs, analysis visits will be represented as follows and in that order:

| Long Name (default) | Short Name |
|---------------------|------------|
| Screening | Scrn |
| Baseline | Base |
| Day 1 | D1 101 |
| Day 8 | D8 |
| Day 29 | D29 |
| Day 43 | D43 |
| Day 57 | D57 |
| Day 209 | D209 |
| Day 394 | D394 |

### **Descriptive Statistics**

If the original data has N decimal places, then the summary statistics will have the following decimal places:

- Minimum, maximum and lower and upper bounds of two-sided 95% CI for percentages: N;
- Mean (including GMT and GMFR), median, lower and upper bounds of two-sided 95% CI for GMT/GMFR: N + 1;
- SD: N + 2.

# **Percentages**

Percentages will be reported to one decimal place. Rounding will be applied, except for percentages < 0.1 but > 0.0 which will be presented as '< 0.1', percentages < 100.0 but > 99.9 which will be presented as '> 99.9' and the percentage equals exactly 100 where it shall be displayed as an integer (100).

Where counts are zero, no percentages will appear in the output.

.ccimal places. Rounding will be applicanted as '< 0.001' and p-values < 1.000 b

.red by the following (unless otherwise indicated in the outless of the property of the state of the policy of the policy o p-values will be reported to three decimal places. Rounding will be applied, except for the p-values < 0.001 which will be presented as '< 0.001' and p-values < 1.000 but > 0.999 which will be presented as '> 0.999'.

Listings
All listing

All listings will be ordered by the following (unless otherwise indicated in the output template):